CLINICAL TRIAL: NCT01700114
Title: Post-Approval Study of MelaFind
Status: Terminated | Type: Observational
Why Stopped: FDA withdrew requirement to complete study
Sponsor: MELA Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol 20111
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Melanoma
Keywords: Pigmented Skin Lesions; Dermatology; Skin Cancer; Melanoma; MelaFind
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pathology slides of biopsied tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MelaFind — The device is used when a dermatologist chooses to obtain additional information on atypical skin lesions for a decision to biopsy.

SUMMARY:
The purpose of this study is to collect data to describe the real-world use and safety and effectiveness of MelaFind® in a post-approval clinical setting.

DETAILED DESCRIPTION:
The primary objective of this study to test the hypothesis that, among eligible and evaluable lesions with central histological reference standard status melanoma or high-grade lesion, the relative sensitivity ρ comparing enrolling dermatologists after MelaFind use with enrolling dermatologists if MelaFind were not available is greater than 110%. This represents a clinically meaningful increase in sensitivity.

The secondary objectives of this study are to evaluate real-world use and safety and effectiveness of MelaFind in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* The lesion is pigmented (i.e., melanin, keratin, blood)
* Clinical management of the lesion by the examining dermatologist is either biopsy of the lesion in toto, or 3-month follow-up of the lesion
* The diameter of the pigmented area is between 2 and 22 millimeters
* The lesion is accessible to the MelaFind hand-held imaging device
* The patient, or a legally authorized representative, has consented to participate in the study and has signed the Informed Consent Form

Exclusion Criteria:

* The patient has a known allergy to isopropyl alcohol
* The lesion has been previously biopsied, excised, or traumatized
* The skin is not intact (e.g., open sores, ulcers, bleeding)
* The lesion is within 1 cm of the eye
* The lesion is on mucosal surfaces (e.g., lips, genitals)
* The lesion is on palmar hands
* The lesion is on plantar feet
* The lesion is on or under nails
* The lesion is located on or in an area of visible scarring
* The lesion contains foreign matter (e.g., tattoo, splinter, marker)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients of any age, race, ethnicity, or gender, presenting with pigmented skin lesions that that meet the Indications for Use and Lesion Inclusion and Exclusion Criteria, including signing the Informed Consent Form, are eligible to participate in this study. This single-arm study has one study group consisting of eligible lesions on eligible patients.
  Up to six clinical sites in the US will participate in this study, one in each of the six states in which MelaFind is commercially available. Some of the sites will be located in urban settings, and some will be located in a suburban or rural setting. At least 50% of the sites will new, i.e., they did not participate in the MelaFind pivotal study. Some sites will be academic centers and some private practices.
Sampling Method: Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Relative sensitivity comparing enrolling dermatologists after MelaFind use with enrolling dermatoligsts if MelaFind were not available | 6 years

SECONDARY OUTCOMES:
To describe characteristics of patients and lesions with MelaFind, the experience of using MelaFind, distribution of test results, and details on biopsied lesions. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Armand Cognetta, MD, Principal Investigator — Dermatology Associates of Tallahassee; Timothy Wang, MD, Principal Investigator — The John's Hopkins University; Meg Gerstenblith, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Robert Nossa, MD, Principal Investigator — The Dermatology Group, P.C; Arthur Sober, MD, Principal Investigator — Massachusetts General Hospital; Joel Cohen, MD, Principal Investigator — AboutSkin Dermatology and DermSurgery
Locations (6):
- United States (6):
  - AboutSkin Dermatology and DermSurgery, Englewood, Colorado
  - Dermatology Associates of Tallahassee, Tallahassee, Florida
  - The Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Dermatology Group, P.C., Verona, New Jersey
  - University Hospitals Case Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No